CLINICAL TRIAL: NCT04786470
Title: Transversus Abdominis Plane Catheter Following Kidney Transplantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Andrew Rasmussen, Kidney and Pancreas Transplantation Fellow, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116618
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Pain, Postoperative; Kidney Transplant
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local Anaesthetic Infusion (Active Comparator)
  Interventions: Drug: Ropivacaine
- Saline Infusion (Sham Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — Ropivacaine infusion via transversus abdominis plane catheter.
  Arms: Local Anaesthetic Infusion
Drug: Saline — Saline infusion via transversus abdominis plane catheter.
  Arms: Saline Infusion

SUMMARY:
Continuous Infusion of Local Anesthetic After Kidney Transplantation

This is a phase III, randomized, double-blinded, sham-controlled trial comparing the use of a continuous infusion of local anesthetic via transversus abdominis plane (TAP) catheter to a saline infusion (sham) via TAP catheter along with standard postoperative analgesia in patients undergoing kidney transplantation. Patients will have a TAP catheter placed at the time of kidney transplantation by the surgical team under direct vision. They are then randomized to a continuous infusion of local anesthetic or saline for 48 hours postoperatively. Both groups will receive a standard postoperative analgesic regimen including a Patient Controlled Analgesic (PCA) pump and multimodal analgesics including acetaminophen and gabapentin.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male, female, non-binary gender, aged >18 years.
4. Undergoing a kidney transplant (deceased or living donor) as treatment for stage 5 chronic kidney disease (Glomerular filtration rate < 15ml/min) either on dialysis, or approaching dialysis
5. No history of allergy to any local anesthetic.
6. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

Exclusion Criteria:

1. Current use of opioid pain medications prior to kidney transplantation.
2. Known allergic reactions to components of any local anesthetic medication.
3. Prior local anesthetic systemic toxicity.
4. History of chronic pain undergoing current active treatment for the same.
5. Age <18 years (this analgesic approach has not been established in this population).
6. Unable or unwilling to use IV PCA pump for any reason (manual dexterity, cognitive impairment, patient choice etc.).
7. Multi-visceral transplantation.
8. Incision other than standard Gibson incision.
9. Unilateral or bilateral nephrectomy at time of kidney transplant.
10. Advanced liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Oral morphine equivalent (OME) | 48 hours post kidney transplantation
  OME in mg

SECONDARY OUTCOMES:
Visual Analog Scale pain rating | 12, 24, and 48 hours post kidney transplantation
  Series of 5 faces that depict discomfort levels ranging from severe pain (score 5) to no pain at all (score 1). The higher the score, the more pain a patient has.
Patient quality of life score | 48 hours post kidney transplantation
Time to return of bowel function postoperatively | Duration of admission
Incidence of local anesthetic systemic toxicity | Duration of admission
Postoperative adverse events (surgical) | Duration of admission
Delayed graft function | Duration of admission
  Defined as the requirement for hemodialysis/peritoneal dialysis within the first 7 days after kidney transplantation for any reason.
Creatinine (mmol/L) at time of discharge | Duration of admission
Length of stay | Duration of admission

IPD SHARING:
Plan to Share IPD: No